CLINICAL TRIAL: NCT00604110
Title: Interest in Biventricular Epicardial Pacing Post Cardiac Surgery in Patients With Left Ventricular Ejection Fractions Less Than 45%
Brief Title: Biventricular Epicardial Pacing Post Cardiac Surgery in Patients With Left Ventricular Ejection Fractions Less Than 45%
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: CHU Clermont-Ferrand, Cardiac surgery center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0028
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure
Keywords: Biventricular pacing; resynchronisation therapy; cardiac surgery; ejection fraction of less 45%
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Other: Biventricular pacing post cardiac surgery — Determine which biventricular pacing after cardiac surgery, in patients with reduced left ventricular function (EF<45%), is hemodynamically favourable.

SUMMARY:
Patients with reduced left ventricular function are at an increased perioperative risk and often need prolonged postoperative treatment on intensive care units. A significant portion of these patients require postoperative pacing. Right ventricular pacing has been shown to be hemodynamically deleterious The aim of this study is to determine which biventricular pacing after cardiac surgery, in patients with reduced left ventricular function (EF≤ 45%), is hemodynamically favourable.

DETAILED DESCRIPTION:
Some patients with left ventricular systolic dysfunction (LVSD) have an inefficient pumping function. These patients have been shown to benefit from a device therapy known as biventricular pacing. Biventricular pacing causes a more coordinated contraction of the heart chambers resulting in improvement in the pumping ability of the heart and blood pressure. Cardiac Resynchronization Therapy (CRT) has established itself as a proven therapy for congestive heart failure in adults, patients showing improvement in exercise tolerance, quality of life, and survival.

In cardiac surgery, a significant number of these patients with left ventricular systolic dysfunction require postoperative pacing. Right ventricular pacing has been shown to be hemodynamically deleterious Whether biventricular pacing in patients with LVSD improves patient outcomes after heart surgery has not been investigated.

The aim of this crossover trial is to compare conventional ventricular pacing and DDD-biventricular in post operative patients with a pre operative ejection fraction less than 45%, in a prospective randomized setting.

We would like to determine whether biventricular pacing optimized by trans thoracic echocardiography of left ventricular, immediately after heart surgery in patients with LVSD will improve the heart function.

Immediately after surgery, the patients will receive atrio ventricular conventional right ventricular pacing, or biventricular pacing depending upon the treatment arm that they were randomized to.

The primary end point is a 15 % improvement in index cardiac measured by thermal dilution and/or echocardiography in intensive care unit.

Furthermore, Plasma N-terminal pro-brain natriuretic peptide (NT-proBNP), cardiac troponin T (cTnT), will be measured in patients undergoing elective cardiac surgery 12 h, 24 h, 48 h and 72 hours after.

This study is important because of a high probability of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Planned CABG and/or valve surgery
* Left ventricular dysfunction (EF≤ 45%)
* Age > 18 years
* able to give written information consent

Exclusion Criteria:

* Existing permanent pace maker
* Atrial fibrillation
* Enrolment in other research protocols
* Inability to give written informed consent
* Heart transplant
* Pre operative cardiovascular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-09 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Determine whether biventricular pacing optimized by trans thoracic echocardiography of left ventricular will improve the heart function | immediately after heart surgery in patients with LVSD

CONTACTS AND LOCATIONS:
Overall Officials: Charles De Riberolles, Pr, Principal Investigator; Stéphane Combes, Dr, Principal Investigator
Locations (1):
- CHU, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Forestier C, Guelon D, Cluytens V, Gillart T, Sirot J, De Champs C. Oral probiotic and prevention of Pseudomonas aeruginosa infections: a randomized, double-blind, placebo-controlled pilot study in intensive care unit patients. Crit Care. 2008;12(3):R69. doi: 10.1186/cc6907. Epub 2008 May 20. PMID 18489775